CLINICAL TRIAL: NCT05613556
Title: Monitoring Physiologic Parameters in Individuals With Diabetic Peripheral Neuropathy: a Prospective Study
Brief Title: Monitoring Physiologic Parameters in Individuals With Diabetic Peripheral Neuropathy
Status: Completed | Type: Observational
Sponsor: Orpyx Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ORPYX
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Diabetic Foot; Diabetic Peripheral Neuropathy
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Orpyx SI® Sensory Insole System — Orpyx SI Sensory Insole System consists of Orpyx Custom Insoles and Orpyx Sensory Technology. The Orpyx Custom Insoles are precisely fabricated for an individual's feet. The Orpyx Sensory Technology, a powered limb overload warning technology, is compatible with the Orpyx Custom Insoles. It is intended for monitoring physiological parameters, such as plantar pressure, motion and temperature, and providing real-time cues for pressure offloading as the patient goes about their daily activities

SUMMARY:
The primary aim of this study is to use the Orpyx® SI Sensory Insole System (Orpyx Medical Technologies Inc., Calgary AB, Canada) ("Orpyx" or "the Company") as an adjunct to diabetic peripheral neuropathy standard of care (SOC), and observe step count, pressure, temperature, and adherence data through remote patient monitoring (RPM). This will provide insights into patient engagement and the benefits of offering remote, preventative care.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed neuropathy and type 1 or 2 diabetes
* Qualification as a "Moderate or High-Risk Participant," as defined by the International Working Group on the Diabetic Foot (IWGDF) Guidelines
* Complete healing of any previous foot ulcers, as defined by complete re-epithelialization of healed ulcer which is confirmed by two medical exams that occur at least two to three weeks apart (V0 and V1)
* Ability to walk independently (without use of wheelchair) for 30 steps
* Aged >18 years
* Ability to understand all the study and device requirements and have a life expectancy greater than the study duration
* 0.6 < [ABI] < 1.2, capillary refill time < 5 seconds (in the last 12 months)
* Subject is willing and able to wear the Orpyx Sensory Insoles and provided diabetic footwear during all weight bearing activities (sitting, standing, walking, and wearing footwear)
* Most recent HbA1c level of < 12.0% (in the last 12 months)
* Subject or caregiver is able to see the bottom of their feet and inspect for redness, callus, and wounds as per standard of care
* Subject is willing to wear the sensory insoles and carry the digital display device all day, but for a minimum of 4.5 hours a day
* Subject is willing to charge the Orpyx SI Sensory Insoles overnight every night

Exclusion Criteria:

* Active ulcer or presence of other open chronic wound (on foot or other body surface), regardless of etiology (e.g., vasculitis, neoplasms, or hematological disorders)
* Past history of known non-neuropathic foot ulcer (i.e., arterial or venous insufficiency ulcer)
* Presence of severe vascular disease (refer to acceptable ABI parameters in section 7.7.1)
* Dementia
* Psychiatric illnesses or social situations that would limit compliance with the study
* Serious underlying balance dysfunction, regardless of etiology
* Significant cardiopulmonary or other systemic disease limiting the participant's ability to walk at least 30 steps or to stand for an amount of time equal to or greater than five (5) minutes
* Current participation in another clinical investigation of a medical device or a drug; or participation in such a study within 30 days prior to this study enrolment
* Current osteomyelitis or gangrene of the lower extremity
* Uncorrected plantar Charcot neuroarthropathy
* Bunion which would predispose ulcer formation (clinician discretion)
* Extreme equinus
* Hallux valgus
* At the start of V1, the subject does not continue to meet the entrance criteria (inclusion and exclusion)
* Hallux rigidus / limitus
* Any condition that would affect or limit the ability to properly fit both shoes with the device under study
* Subject has a history of intercurrent illness or conditions that would compromise the safety of the subject or their ability to participate in this study
* Subject is in a site of care that is not conducive to ambulation or qualify for remote patient care (skilled nursing facility, acute care facility)
* Amputations on the foot which require additive insole modifications (including but not limited to transmetatarsal, toe or ray amputations which create the need for a toe filler, or which prevent the subject from wearing the prescribed footwear)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participant population to be studied will be subjects 18 years of age or older who have been diagnosed with diabetes (Type I or Type II) and neuropathy and who are at moderate to high risk of foot ulceration based on the International Working Group on the Diabetic Foot (IWDGF) guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Frequency and location of high-pressure plantar areas | 3 months
  frequency and location of high-pressure plantar areas

CONTACTS AND LOCATIONS:
Locations (1):
- WAFL Inc / Cutting Edge Research, Circleville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No